CLINICAL TRIAL: NCT03599505
Title: Intraoperative Ultrasonographic Localization of Pulmonary Nodules in Video-assisted Thoracoscopic Surgery
Brief Title: Intraoperative Ultrasonographic Localization of Pulmonary Nodules in VATS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Lei, Chief physician, Shanghai Chest Hospital
Other Study IDs: Chest008
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Ultrasonography
Keywords: intraoperative ultrasonographic localization; pulmonary nodules; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: localization group — Intraoperative ultrasonographic localization will be performed using an ultrasound system (HI VISON Ascendus), which is equipped with a 5-10MHz mechanical probe (EUP-OL531). The accuracy rate of localization will be evaluated using gray scale mode and elastography mode.

SUMMARY:
This study is conducted to explore the feasibility and value of Intraoperative ultrasonographic localization of pulmonary nodules in video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
The study is designed as a single center prospective trial. The participating center is Department of Ultrasound, Shanghai Chest Hospital, Shanghai Jiao Tong University, China. The study is expected to enroll 200 patients. The feasibility and value of Intraoperative ultrasonographic localization of pulmonary nodules in VATS will be explored. The accuracy rate of localization will be evaluated using gray scale mode and elastography mode. Intraoperative ultrasonographic localization will be performed using an ultrasound system (HI VISON Ascendus), which is equipped with a 5-10MHz mechanical probe (EUP-OL531).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are older than 18 year-old.
2. Chest CT shows pulmonary nodule suspected to be malignant that need to undergo VATS.
3. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Patient with severe asthma and pulmonary fibrosis.
2. Refusal of participation.
3. Severe cardiopulmonary dysfunction and other indications that can't receive VATS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 year-old with chest CT showing pulmonary nodule that need to undergo VATS will be enrolled in the study. Patient with severe cardiopulmonary dysfunction and other indications that can't receive VATS will be excluded.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy rate of localization | one year
  The accuracy rate of localization will be evaluated using gray scale mode and elastography mode using pathology as a reference.

SECONDARY OUTCOMES:
Correlation of lesion size and localization | one year
  Whether lesion size affects localization will be explored in the study.
Correlation of distance between the lesion and pleura and localization | one year
  Whether distance between the lesion and pleura affects localization will be explored.
Time of localization | one week
  The time of intraoperative ultrasonographic localization will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, MD, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kondo R, Yoshida K, Hamanaka K, Hashizume M, Ushiyama T, Hyogotani A, Kurai M, Kawakami S, Fukushima M, Amano J. Intraoperative ultrasonographic localization of pulmonary ground-glass opacities. J Thorac Cardiovasc Surg. 2009 Oct;138(4):837-42. doi: 10.1016/j.jtcvs.2009.02.002. Epub 2009 Mar 26. PMID 19660350
- [Background] Mattioli S, D'Ovidio F, Daddi N, Ferruzzi L, Pilotti V, Ruffato A, Bolzani R, Gavelli G. Transthoracic endosonography for the intraoperative localization of lung nodules. Ann Thorac Surg. 2005 Feb;79(2):443-9; discussion 443-9. doi: 10.1016/j.athoracsur.2004.07.087. PMID 15680811
- [Background] Nakashima S, Watanabe A, Obama T, Yamada G, Takahashi H, Higami T. Need for preoperative computed tomography-guided localization in video-assisted thoracoscopic surgery pulmonary resections of metastatic pulmonary nodules. Ann Thorac Surg. 2010 Jan;89(1):212-8. doi: 10.1016/j.athoracsur.2009.09.075. PMID 20103238
- [Background] Pittet O, Christodoulou M, Pezzetta E, Schmidt S, Schnyder P, Ris HB. Video-assisted thoracoscopic resection of a small pulmonary nodule after computed tomography-guided localization with a hook-wire system. Experience in 45 consecutive patients. World J Surg. 2007 Mar;31(3):575-8. doi: 10.1007/s00268-006-0343-7. PMID 17318707
- [Background] Chen W, Chen L, Yang S, Chen Z, Qian G, Zhang S, Jing J. A novel technique for localization of small pulmonary nodules. Chest. 2007 May;131(5):1526-31. doi: 10.1378/chest.06-1017. PMID 17494801